CLINICAL TRIAL: NCT01493830
Title: Proposed Studies on the Role of Growth Factor Receptor Trafficking in Neuroblastoma Pathogenesis
Brief Title: Biomarkers in Tumor Samples From Younger Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL12B4; COG-ANBL12B4 (Other: Children's Oncology Group); NCI-2012-00091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL12B4 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — In Situ Hybridization, Fluorescence; Gene Expression Profiling; Microarray Analysis; Immunohistochemistry; Microscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: protein analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: microscopy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in tumor samples from younger patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the expression of UBE4B, hrs, and members of the ubiquitination protein complex in previously banked primary neuroblastoma tumor samples from the Children's Oncology Group.
* To determine the correlation of expression levels and cellular localization of the UBE4B and hrs proteins with growth factor-receptor tumor cell-surface expression.
* To determine the 1p36 deletion status by fluorescence in situ hybridization (FISH) analysis and their association with expression levels of UBE4B and hrs in previously banked primary neuroblastoma tumor samples from the Children's Oncology Group.

OUTLINE: Banked tumor tissue samples are analyzed for expression of UBE4B, hrs, members of the ubiquitination protein complex, growth factor receptors, and 1p36 deletion status by immunohistochemistry (IHC), fluorescent microscopy, and fluorescence in situ hybridization (FISH).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor tissue microarrays from the Children's Oncology Group neuroblastoma tumor bank

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Expression of UBE4B, hrs, and members of the ubiquitination protein complex
Expression levels and cellular localization of the UBE4B, hrs, and growth factor receptors
1p36 deletion status and its association with UBE4B

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zage, MD, PhD, Principal Investigator — Texas Children's Cancer Center